CLINICAL TRIAL: NCT07207148
Title: People With Multiple Sclerosis Treated With Ocrelizumab and GLP-1 Agonists
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Farrah Mateen, Professor of Neurology, Northwestern University Feinberg School of Medicine
Other Study IDs: STU00224018
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Ocrelizumab; GLP-1; Obesity; Weight loss; Progressive MS; Multiple sclerosis; Biomarkers; Weight; Overweight; Neuroprotection; Semaglutide; glucagon-like peptide-1
MeSH Terms: conditions — Multiple Sclerosis; Obesity; Weight Loss; Body Weight; Overweight | interventions — Glucagon-Like Peptide 1; ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Aim 1: The cohort will implement patient-reported outcome measures (PROMs) in 60 people with MS already treated with both Ocrelizumab and a GLP-1 agonist to assess progression and ambulation, while recording drug tolerability and potential adverse events, weight loss, disease-based outcomes focused on progression, and MS-focused quality of life.
  Interventions: Drug: GLP-1; Drug: Ocrelizumab (US)
- Aim 2: The cohort will include a single-arm, open-label trial of 40 Ocrelizumab-treated MS patients who are soon starting GLP-1 agonists, monitored prospectively for 2 years to measure MS progression (clinical disability worsening, stability or improvement) every 3 months, including (a) clinical assessments (e.g. EDSS, 25-foot timed walk, SDMT) as used in the ORATORIO trial of Ocrelizumab, (b) PROMs on progression in MS including fatigue, ambulation distance, mood; and (3) simple objective biomarkers of disease (e.g. plasma neurofilament light chain, glial fibrillary acidic protein).
  Interventions: Drug: GLP-1; Drug: Ocrelizumab (US)

INTERVENTIONS:
Drug: GLP-1 — Glucagon-like peptide-1 agonist agent is the study agent of interest. This study will not supply the GLP-1 drug but depends on the patient's clinical prescription of this drug.
  Other Names: Glucagon-like peptide-1; GLP-1 Agonist
Drug: Ocrelizumab (US) — All participants will be treated with Ocrelizumab for the indication of MS; however, the study will not provide Ocrelizumab as it will be part of the participant's routine clinical care.
  Other Names: Ocrevus

SUMMARY:
The primary outcome measure is PIRA (progression independent of relapse activity), based primarily on clinical assessment, dichotomized as present or not.

For Aim 1, the cohort, patient-derived disability status (PDDS) score, and ambulation score (self-reported) will be the primary endpoints of interest.

For Aim 2, the clinical trial, PIRA will be measured pre-GLP-1 start and at study end (week 72). A composite score of disability, similar to the ORATORIO13 trial will be constructed including EDSS score, 25-foot timed walk, 9-hole peg test, and SDMT score.

DETAILED DESCRIPTION:
STUDY PROCEDURES:

Aim 1 will allow fully remote participation, drawing from geographically diverse settings throughout the USA. Participants in Aim 1 do not need to visit the study site in person or be independently mobile but must be continuously available during the study timeframe remotely for PROMS and study surveys and calls.

Participants will be enrolled for an estimated 72 weeks: Measurements will be requested every four weeks (i.e. q28 days) on a specifically designed survey instrument for MS participants. Participants will be asked to report medication dosing, adherence to medicine, tolerability, weight, height, and exercise activities. Self-reported scales will be administered to the participants as well (measuring disability, fatigue, mood, and quality of life).

Participants must be currently on Ocrelizumab (last dose within the past <6 months) and currently taking a GLP-1 medication.

Participants will be contacted and interviewed via Zoom every 6 months to ensure study procedures are going as planned, verify data reported on medication and MS disease history, and ensure study procedures are operating smoothly. Participants who do not complete the surveys within 7 days of the scheduled timing will be contacted by a study coordinator by phone up to 3 times. Participants will also be asked to report any medication changes, dose changes, or discontinuations if they occur at any point between study visits.

Participants will be enrolled until a total of 40 individual participants are reached. Study procedures for each group are listed in Tables 1 and 2. All scheduled events will be part of the study and not part of routine clinical care.

Allocation and Blinding

All participants will be treated with the two drugs of interest: Ocrelizumab and the GLP-1 agonist. The participants will be blinded to the study outcome of interest, i.e. progression or PIRA. The investigators will not be blinded to the study outcome. The participants will not have access to their prior PDDS scores on file, earlier in the study. The EDSS raters will not have access to the prior EDSS scores on file, earlier in the study. The statisticians will not be blinded to the study outcome.

Criteria for Study Drug Discontinuation in a Single Participant

Reasons for GLP-1 agonist drug discontinuation will be at the discretion of the treating prescriber include: (1) laboratory test abnormalities (e.g. transaminitis) whether related to the drugs or not; (2) intercurrent illness; (3) severe intolerance to the GLP-1 agonist; (4) lack of access to the GLP-1 drug within an affordable range; (5) patient preference; (6) achieved weight target earlier than anticipated; or (7) any other reason as determined by the prescribing physician or study principal investigator.

Criteria for Study Withdrawal of a Participant

Participants who discontinue GLP-1 agonist drugs for any reason, including tolerability, cost, desired weight loss outcome, etc., will continue to be observed until the end of the study period. It is possible that participants will have periods of discontinuation and then resume GLP-1 agonist treatment. The participant will be observed until (a) week 72 visit (i.e. end of study period), (b) participant withdrawal with no consent to continue monitoring, or (c) investigator-decided withdrawal of a participant from the study (e.g. severe medical illness preventing study completion, departure far from study site, etc.).

There is no anticipated drug development or future product anticipated in this study. A study participant will not have any right to compensation or ownership interest related to such development.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS (2019 revised McDonald criteria) of any type (PPMS, RRMS, SPMS) by a neurologist,
* Adult age 18-70 years,
* BMI >=24.0 kg/m2,
* Taken at least one dose of Ocrelizumab prior to study entry,
* EDSS <7.0,
* Able to provide individual informed consent,
* MRI available to confirm the diagnosis of MS.

Exclusion Criteria:

* Prior exposure to Mavenclad, Lemtrada, Cyclophosphamide, stem cell transplant or related bone marrow suppressive treatment,
* Current clinical trial participant,
* Unable to speak a language for which translation can be found in the hospital system,
* Unclear documentation of MS diagnosis or prior or current MS treatment,
* Relapse within the past 3 months,
* Recent major surgical procedure in the past 6 months,
* Exposure to steroids (systemic) within the past 3 months,
* Not on Ocrelizumab in the past >9 months,
* Moribund status,
* Underweight or experiencing protein malnutrition,
* Unable to provide consent voluntarily due to reasons of capacity or other reasons (e.g. incarcerated, dementia, etc.),
* Unable to complete the study activities for any reason as deemed by the study investigator.

Additional Inclusion Criteria Aim 1:

* Exposed to GLP-1 agonist treatment in the last 3 years or less, or starting on a GLP-1 agonist in the coming <3 months,
* Willing to report monthly patient-reported outcomes remotely or in-person.

Additional Inclusion Criteria Aim 2:

* Able to present for baseline and follow up in person,
* Unexposed to a GLP-1 agonist in the past year,
* Starting on a GLP-1 agonist in the next <6 months,
* Plan to be exposed to GLP-1 agonist for a minimum of 72 weeks following enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with multiple sclerosis already treated with both Ocrelizumab and are either currently on a GLP-1 agonist or who are soon starting a GLP-1 agonist.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
PIRA | From enrollment to the end of study at 72 weeks.
  The primary outcome measure is PIRA (progression independent of relapse activity), based primarily on clinical assessment, dichotomized as present or not.

SECONDARY OUTCOMES:
Neurofilament light chain | From the start of Aim 2 to the end of treatment at 72 weeks.
  There will be blood draws in Aim 2's clinical trial population. Aim 1's observational, interactive cohort will have an optional blood draw component. In both cases, the blood tests will involve send out testing for neurofilament light chain and in Aim 2, glial fibrillary acidic protein.

CONTACTS AND LOCATIONS:
Overall Officials: Farrah J Mateen, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharrad D, Chugh P, Slee M, Bacchi S. Defining progression independent of relapse activity (PIRA) in adult patients with relapsing multiple sclerosis: A systematic review✰. Mult Scler Relat Disord. 2023 Oct;78:104899. doi: 10.1016/j.msard.2023.104899. Epub 2023 Jul 20. PMID 37499338
- [Background] Montalban X, Hauser SL, Kappos L, Arnold DL, Bar-Or A, Comi G, de Seze J, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Rammohan KW, Selmaj K, Traboulsee A, Sauter A, Masterman D, Fontoura P, Belachew S, Garren H, Mairon N, Chin P, Wolinsky JS; ORATORIO Clinical Investigators. Ocrelizumab versus Placebo in Primary Progressive Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):209-220. doi: 10.1056/NEJMoa1606468. Epub 2016 Dec 21. PMID 28002688
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Diz-Chaves Y, Maastor Z, Spuch C, Lamas JA, Gonzalez-Matias LC, Mallo F. Glucagon-like peptide 1 receptor activation: anti-inflammatory effects in the brain. Neural Regen Res. 2024 Aug 1;19(8):1671-1677. doi: 10.4103/1673-5374.389626. Epub 2023 Dec 11. PMID 38103230
- [Background] Sadek MA, Kandil EA, El Sayed NS, Sayed HM, Rabie MA. Semaglutide, a novel glucagon-like peptide-1 agonist, amends experimental autoimmune encephalomyelitis-induced multiple sclerosis in mice: Involvement of the PI3K/Akt/GSK-3beta pathway. Int Immunopharmacol. 2023 Feb;115:109647. doi: 10.1016/j.intimp.2022.109647. Epub 2022 Dec 28. PMID 36584570
- [Background] Udawatta M, Fidalgo N, Mateen FJ. Multiple sclerosis patients taking glucagon-like peptide-1 receptor (GLP-1) agonists: a single-institution retrospective cohort study of tolerability and weight loss. Neurol Sci. 2025 Jan;46(1):343-349. doi: 10.1007/s10072-024-07701-7. Epub 2024 Jul 20. PMID 39030327
- [Background] Li M, Lin H, Yang Q, Zhang X, Zhou Q, Shi J, Ge F. Glucagon-like peptide-1 receptor agonists for the treatment of obstructive sleep apnea: a meta-analysis. Sleep. 2025 Apr 11;48(4):zsae280. doi: 10.1093/sleep/zsae280. PMID 39626095
- [Background] Meissner WG, Remy P, Giordana C, Maltete D, Derkinderen P, Houeto JL, Anheim M, Benatru I, Boraud T, Brefel-Courbon C, Carriere N, Catala H, Colin O, Corvol JC, Damier P, Dellapina E, Devos D, Drapier S, Fabbri M, Ferrier V, Foubert-Samier A, Frismand-Kryloff S, Georget A, Germain C, Grimaldi S, Hardy C, Hopes L, Krystkowiak P, Laurens B, Lefaucheur R, Mariani LL, Marques A, Marse C, Ory-Magne F, Rigalleau V, Salhi H, Saubion A, Stott SRW, Thalamas C, Thiriez C, Tir M, Wyse RK, Benard A, Rascol O; LIXIPARK Study Group. Trial of Lixisenatide in Early Parkinson's Disease. N Engl J Med. 2024 Apr 4;390(13):1176-1185. doi: 10.1056/NEJMoa2312323. PMID 38598572
- [Background] Lincoff AM, Brown-Frandsen K, Colhoun HM, Deanfield J, Emerson SS, Esbjerg S, Hardt-Lindberg S, Hovingh GK, Kahn SE, Kushner RF, Lingvay I, Oral TK, Michelsen MM, Plutzky J, Tornoe CW, Ryan DH; SELECT Trial Investigators. Semaglutide and Cardiovascular Outcomes in Obesity without Diabetes. N Engl J Med. 2023 Dec 14;389(24):2221-2232. doi: 10.1056/NEJMoa2307563. Epub 2023 Nov 11. PMID 37952131
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Background] Fitzgerald KC, Salter A, Tyry T, Fox RJ, Cutter G, Marrie RA. Measures of general and abdominal obesity and disability severity in a large population of people with multiple sclerosis. Mult Scler. 2020 Jul;26(8):976-986. doi: 10.1177/1352458519845836. Epub 2019 May 13. PMID 31079537
- [Background] Hedstrom AK, Brenner N, Butt J, Hillert J, Waterboer T, Olsson T, Alfredsson L. Overweight/obesity in young adulthood interacts with aspects of EBV infection in MS etiology. Neurol Neuroimmunol Neuroinflamm. 2020 Dec 15;8(1):e912. doi: 10.1212/NXI.0000000000000912. Print 2021 Jan. PMID 33465039
- [Background] Mandato C, Colucci A, Lanzillo R, Staiano A, Scarpato E, Schiavo L, Operto FF, Serra MR, Di Monaco C, Napoli JS, Massa G, Vajro P. Multiple Sclerosis-Related Dietary and Nutritional Issues: An Updated Scoping Review with a Focus on Pediatrics. Children (Basel). 2023 Jun 7;10(6):1022. doi: 10.3390/children10061022. PMID 37371254
- [Background] Lutfullin I, Eveslage M, Bittner S, Antony G, Flaskamp M, Luessi F, Salmen A, Gisevius B, Klotz L, Korsukewitz C, Berthele A, Groppa S, Then Bergh F, Wildemann B, Bayas A, Tumani H, Meuth SG, Trebst C, Zettl UK, Paul F, Heesen C, Kuempfel T, Gold R, Hemmer B, Zipp F, Wiendl H, Lunemann JD; German Competence Network Multiple Sclerosis (KKNMS). Association of obesity with disease outcome in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2023 Jan;94(1):57-61. doi: 10.1136/jnnp-2022-329685. Epub 2022 Nov 1. PMID 36319190

DOCUMENTS (2):
  • Study Protocol (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT07207148/Prot_000.pdf
  • Informed Consent Form (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT07207148/ICF_001.pdf